CLINICAL TRIAL: NCT06839547
Title: A Prospective, Multicenter, Observational Cohort Study to Evaluate the Efficacy and Safety of a Novel Anti-tumor Drug As a Radiosensitizer in Patients with Advanced Breast Cancer Brain Metastasis.
Status: Not yet recruiting | Type: Observational
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Ma Fei，MD, Deputy Director of the Department of Medical Oncology, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Other Study IDs: NCC5104
Record Dates: First submitted 2025-02-18; First posted 2025-02-21 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2024-09

CONDITIONS: Advanced Breast Cancer Brain Metastasis
MeSH Terms: interventions — Radiotherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — Peripheral blood and tissue samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Radiotherapy + Novel Anti-tumor Drug — 1. Novel anti-tumor drugs [including: ADC drugs (such as T-DXd, T-DM1, etc.), CDK4/6 inhibitors, TKI drugs (such as Pyrotinib, Tucatinib, etc.), novel chemotherapy drugs (such as Utidelone, Irinotecan liposomes, etc.), Bevacizumab, PD-1/PD-L1 inhibitors, etc.]
  2. Radiotherapy

SUMMARY:
A prospective, multicenter, observational cohort study to evaluate the efficacy and safety of a novel anti-tumor drug as a radiosensitizer in patients with advanced breast cancer brain metastasis.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females who are at least 18 years of age on the day of signing the informed consent form.
2. Patients with advanced breast cancer that is inoperable and has metastasized to the brain, confirmed by histology or cytology.
3. Patients who are planned to receive, currently receiving, or have completed intracranial radiotherapy after discussion by a multidisciplinary team (MDT) at the stage of brain metastasis.
4. Patients who are planned or currently receiving a systemic treatment regimen with a novel anti-tumor drug selected by the physician, within 3 weeks before radiotherapy, during radiotherapy, or within 3 weeks after completion of radiotherapy. These drugs include:

   ADC drugs (such as T-DXd, T-DM1, etc.), CDK4/6 inhibitors, TKI drugs (such as Pyrotinib, Tucatinib, etc.), Novel chemotherapy drugs (such as Utidelone, Irinotecan liposomes, etc.), Bevacizumab, PD-1/PD-L1 inhibitors, etc.
5. Patients with a traceable medical history during the treatment period.
6. Patients who are able to sign the informed consent form to participate in the study.

Exclusion Criteria:

1. The subject has leptomeningeal metastasis.
2. If the patient has concurrent brain metastasis, the neurological symptoms are too severe to cooperate with radiotherapy.
3. The subject has not signed the informed consent form.
4. Pregnant or breastfeeding women.
5. Other situations deemed by the investigator as unsuitable for inclusion in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study plans to enroll 100 subjects with breast cancer brain metastasis. These subjects have been assessed by a multidisciplinary team (MDT) and are planned to receive or have already received intracranial radiotherapy. They are also planned to receive or are currently receiving treatment with novel anti-tumor drugs [including: ADC drugs (such as T-DXd, T-DM1, etc.), CDK4/6 inhibitors, TKI drugs (such as Pyrotinib, Tucatinib, etc.), novel chemotherapy drugs (such as Utidelone, Irinotecan liposomes, etc.), Bevacizumab, PD-1/PD-L1 inhibitors, etc.].
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2028-09-10 (Estimated); Study Completion 2028-09-10 (Estimated)

PRIMARY OUTCOMES:
Intracranial Progression-Free Survival | 24 months
  The time from the randomization of the subject to the first documented tumor progression (PD) or death due to any cause.